CLINICAL TRIAL: NCT05219318
Title: SPICI: Strategic Treatment Pause of First-line Immune Check Point Inhibitor + VEGFR-Tyrosine Kinase Inhibitor in Good or Only One Adverse Prognostic Factor in Intermediate Risk Metastatic Renal Cell Carcinoma (mRCC) With an Objective Response: a Randomised, Non-inferiority Phase III Study
Brief Title: Treatment Pause Versus Treatment Continuation in IMDC Good or Intermediate Risk With Only One Adverse Prognostic Factor in mRCC Patients With an Objective Response at 12 Months of Treatment With PD1/ PDL1 ICIs + VEGFR-Tyrosine Kinase Inhibitors
Acronym: SPICI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2021/08
Record Dates: First submitted 2022-01-20; First posted 2022-02-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Renal Cell Carcinoma; Good or Only One Adverse Prognostic Factor Intermediate Risk Per IMDC Score
Keywords: Metastatic renal cell carcinoma (mRCC); Objective response; Treatment pause; Treatment continuation
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment pause (Experimental): Treatment pause for 12 months
  Interventions: Other: Treatment pause
- Treatment continuation (Active Comparator): Treatment continuation regimens with PD-1/PD-L1 ICI + VEGFR-TKI until disease progression or unacceptable toxicity
  Interventions: Drug: Combination PD-1/PD-L1 ICI + VEGFR-TKI

INTERVENTIONS:
Drug: Combination PD-1/PD-L1 ICI + VEGFR-TKI — The study will enroll patients achieving an objective response beween the end of the 11th month and the end of the 13th month of treatment with the combination PD-1/PD-L1 ICI + VEGFR-TKI as recommended in the Summary of Product Characteristics (SmPC)
  Arms: Treatment continuation
Other: Treatment pause — Combination regimens discontinuation until progression with the possibility to resume initial combination regimens at progression
  Arms: Treatment pause

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of treatment pause versus treatment continuation in good or intermediate risk with only one adverse prognostic factor as per IMDC mRCC patients with a confirmed objective response between the end of the 11th month to th end of the 13th month of treatment with PD-1/PD-L1 ICI plus VEGFR-TKI.

Tolerance and quality of life of treatment pause with PD-1/PD-L1 ICI + VEGFR-TKI compared to treatment continuation will be reported. In France, its impact on healthcare resource utilization will also be assessed.

DETAILED DESCRIPTION:
Although multiple combinations therapies in particular PD-1/PD-L1 immune-checkpoint inhibitors (PD-1/PD-L1 ICIs) in combination with vascular endothelial growth factor receptor tyrosine kinase inhibitors (VEGFR-TKIs) are approved and have improved patient's outcomes with mRCC, they are maintained until disease progression and treatment pause after an objective response has not been fully explored [5-7]. The good-risk population is characterised by prolonged survival therefore a treatment pause in this population could impact the quality of life, safety and total cost of care, without impacting outcome. As well, intermediate risk population group is heterogeneous, while the one's with only one adverse prognostic factor seems to be closed to the outcome of good risk population [11-15]. As the purpose of the study is to target patients with an objective response, there is already a selection of patients with a better outcome.

Patient will be randomised after 11 to 13 months of treatment with PD-1/PD-L1 ICI plus VEGFR-TKI (treatment pause versus treatment continuation) and follow every 3 months for a period of 12 months following by 12 additional months for survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing informed consent form
* Signed informed consent form
* Histological confirmation of RCC with a Clear-cell component, including subject who also have a sarcomatoïd feature
* Advanced (not amenable to curative surgery or radiation therapy) or Metastatic RCC (American Joint Committee on Cancer [AJCC] Stage IV)
* Participants with good or intermediate risk with only one adverse prognostic factor will be eligible as per International Metastatic RCC Database Consortium (IMDC) criteria
* Prior first line therapy for mRCC with the combination of PD-1/ PD-L1 ICI plus VEGFR-TKI
* First line treatment with the combination of PD-1/PD-L1 ICI and VEGFR-TKI must be ongoing whatever the dose with no period of discontinuation > 6 consecutive weeks during treatment of the PD-1/PD-L1 ICI, and 2 consecutive weeks in the last 3 months before randomisation for the VEGFR-TKI
* Patients with an objective response (complete response or partial response) between the end of 11th month and the end of the 13th month of the combination treatment with PD-1/PD-L1 ICI and VEGFR-TKI. CT scan at the initiation of this treatment must be available.
* Karnofsky Performance Status (KPS) grade ≥ 70%
* Measurable disease as per RECIST v1.1 per investigator on CT scan at the initiation of first line treatment with combination treatment with PD-1/PD-L1 ICI and VEGFR-TKI
* Adequate organ function
* Females of childbearing potential must use a highly effective contraception (combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral ; intravaginal ;transdermal) ; progestogen-only hormonal contraception associated with inhibition of ovulation (oral ; injectable ; implantable ; intrauterine device (IUD) ; intrauterine hormone-releasing system ( IUS)) ; bilateral tubal occlusion ; vasectomised partner ; sexual abstinence) and continue its use for 5 months after the last PD1/PD L1 ICI administration.
* Sexually active male patients must agree to use condoms and continue its use for 5 months after the last PD1/PD L1 ICI administration.
* Willingness and ability to comply with study procedures.
* Patient affiliated to a social security system or benefit from the same system

Exclusion Criteria:

* Prior therapy with PD-1/PD-L1 ICI or VEGFR-TKI monotherapy.
* Poorly controlled hypertension despite antihypertensive therapy
* More than one adverse prognostic factor (IMDC criteria)
* Women who are pregnant or lactating;
* Current participation in an investigational program
* Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study
* Adults who are the subject of legal protection measures
* Persons deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants without progression | Up to 12 months after randomisation
  Disease progression at up to 12 months after randomisation will be based on a blinded independent central review (BICR) according to RECIST v1.1 criteria, with tumor assessment performed every 12 weeks during study participation

SECONDARY OUTCOMES:
Overall safety profile and tolerability event | Up to 12 months after randomisation
  Proportion of participants who experience an adverse event or serious adverse event and mean number of adverse events or serious adverse events up to 12 months after randomisation
Overall survival (OS) | From randomisation until 2 years of follow-up
  OS is defined as the time between the date of randomisation and the date of death due to any cause
Progression-free survival (PFS) | From randomisation until 2 years of follow-up
  PFS is defined as the time between date of randomisation and the first date of the documented disease progression, or death due to any cause, whichever occurs first
Mean change in quality of life | Up to 12 months after randomisation
  Measured by the NCCN functional assessment of cancer therapy-kidney symptom index (FKSI-19). The NCCN FKSI-19 is a 19-item scale that measures tumor specific health-related quality of life in kidney cancer participants. A higher score indicates fewer symptoms
Quality-adjusted survival | Up to 12 months after randomisation
  The quality-adjusted time without symptoms or toxicity (Q-TWiST) is a simultaneous assessment of time without toxicity or disease progression, which essentially examines the trade-off between AEs and treatment benefits
Anxiety and depression | Up to 12 months after randomisation
  Mean scores in the Hospital Anxiety and Depression Scale at up to 12 months after randomisation
Site and distribution of the sites of progression: known lesions, new lesion(s) or both | From randomisation until 2 years of follow-up
Distribution of treatment modality after progression | From randomisation until 2 years of follow-up
  Proportion of participants treated after progression with surveillance, focal treatment or general treatment
Percentage of patients with status SD or in objective response at 6 months after restarting PD-1/PD-L1 ICI + VEGFR-TKI | From randomisation until 2 years of follow-up
Healthcare resource utilisation | Up to 12 months after randomisation
  Costs of care will be estimated in the perspective of the French Healthcare System over a 12-month times horizon. Conventional tariffs of hospitalizations will be used to calculate costs

CONTACTS AND LOCATIONS:
Overall Officials: Marine GROSS-GOUPIL, MD PhD, Principal Investigator — University Hospital, Bordeaux
Locations (26):
- France (26):
  - CH de la Cote Basque - Service d'Oncologie, Bayonne
  - CHU de Bordeaux - Service d'Oncologie, Bordeaux
  - Centre François Baclesse - Service d'Oncologie, Caen
  - Centre Jean Perrin - Service d'Oncologie, Clermont-Ferrand
  - AP-HP - Henri Mondor - Service d'Oncologie, Créteil
  - Centre Georges-François Leclerc - Service d'Oncologie, Dijon
  - CHU Grenoble Alpes - Service d'Oncologie, Grenoble
  - CHU de Limoges - Service d'Oncologie, Limoges
  - Polyclinique de Limoges - Service d'Oncologie, Limoges
  - Centre Leon Berard - Service d'Oncologie, Lyon
  - Hospices Civils de Lyon - Service d'Oncologie, Lyon
  - Institut Paoli-Calmettes - Service d'Oncologie, Marseille
  - Institut Régional du Cancer - Service d'Oncologie, Montpellier
  - Centre Antoine Lacassagne - Service d'Oncologie, Nice
  - AP-HP - Hôpital Européen Georges Pompidou - Service d'Oncologie, Paris
  - AP-HP - Hôpital Saint Louis - Service d'Oncologie, Paris
  - CHU de Poitiers - Service d'Oncologie, Poitiers
  - Centre Eugène Marquis - Service d'Oncologie, Rennes
  - CHU de Saint-Etienne - Service d'Oncologie, Saint-Etienne
  - CHU de la Réunion Site Sud - Service d'Oncologie, Saint-Pierre
  - Institut de cancérologie Strasbourg Europe - Service d'Oncologie, Strasbourg
  - Hopital Foch - Service d'Oncologie, Suresnes
  - IUCT Oncopole - Service d'Oncologie, Toulouse
  - CHU de Tours - Service d'Oncologie, Tours
  - Institut de Cancérologie de Lorraine - Service d'Oncologie, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy - Service d'Oncologie, Villejuif